CLINICAL TRIAL: NCT05573282
Title: Observation Study of Sequential Regorafenib Combined With Immunocheckpoint Inhibitors After Hepatic Artery Infusion Chemotherapy for Advanced Hepatocellular Carcinoma
Brief Title: Observation Study of Sequential Regorafenib Plus ICIs After HAIC for Advanced Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Zhao, Professor, Sun Yat-sen University
Other Study IDs: B2022-334-01
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic arterial infusion chemotherapy; Regorafenib; Immunocheckpoint inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sequential therapy of Regorafenib combined with ICIs: Sequential therapy of Regorafenib combined with one kind of ICIs after standard HAIC treatment in advanced hepatocellular carcinoma (HCC).
  ICIs: atezolizumab, pembrolizumab, nivolumab, camrelizumab, tislelizumab, sintilimab or other ICIs.
  Interventions: Other: Regorafenib combine with ICIs

INTERVENTIONS:
Other: Regorafenib combine with ICIs — Regorafenib: 80mg/day, PO, QD, d1～d21, Q4W ICIs: 200mg/day, IV, d1,Q3W

SUMMARY:
Hepatic artery infusion chemotherapy (HAIC) has shown promising outcomes in patients with advanced hepatocellular carcinoma (HCC). Some patients can be converted to loco-regional therapies after 4-6 cycles of HAIC treatment. But most of these patients still need to concern the sequential treatment after standard HAIC treatment (4-6 cycles). Combination of anti-angiogenic molecular targeted therapy and immune checkpoint inhibitor (ICI) therapy has shown promising antitumor activity in HCC. Regorafenib is one of the standard second-line systemic therapy for advanced HCC. In this study, we will evaluate the efficacy and safety of sequential therapies of Regorafenib plus ICI in patients with advanced HCC who have completed 4-6 cycles of HAIC.

DETAILED DESCRIPTION:
The standard procedure for HAIC is that femoral artery puncture and catheterization are performed in every cycle of treatment, a micro-catheter is inserted and located in feeding hepatic artery. The therapeutic scheme is modified FOLFOX6 regimens including oxaliplatin, leucovorin and Fluorouracil. All chemo-drugs are given by HAI. A total of 4-6 cycles of HAIC are performed and the treated efficacy is evaluated. Patient who is not suitable for loco-regional therapies after 4-6cycles of HAIC becomes to the candidate of sequential therapies of regorafenib plus ICIs. The regorafenib 80 mg/day was uses in sequential treatment. And ICIs were used intravenously at the standard dose. Patients received sequential treatment will begin no earlier than 30 days following the last HAIC procedure.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent must be obtained prior to any screening procedures.

* Cytohistological confirmation is required for diagnosis of HCC.
* Patients with advanced (unresectable and/or metastatic, stage C based on Barcelona-Clinic Liver Cancer [BCLC] staging classification) hepatocellular carcinoma who have completed 4-6 cycles HAIC. Treated efficacy evaluation has confirmed that these patients are not suitable for loco-regional therapies or surgical resection.
* At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1. Lesions previously treated with local therapy, such as radiation therapy, hepatic arterial embolization, radiofrequency ablation, and percutaneous interventional therapy should not be selected unless progression is noted at baseline, in which case, these lesions would be considered as non-target lesions.
* Current cirrhotic status of Child-Pugh class A-B, with no encephalopathy. Ascites controlled by diuretics is permitted in this study.
* Availability of a representative tumor tissue specimen (archival tumor tissue is allowed) at pre-screening.
* Eastern Cooperative Oncology Group Scale for Assessment of Patient Performance Status ≤ 2.
* Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 4 weeks after the completion of trial.
* Adequate bone marrow, liver and renal function as assessed by central lab by means of the following laboratory requirements from samples within 7 days prior to procedure:
* Hemoglobin > 100g/L
* Absolute neutrophil count >3.0 ×109/L
* Neutrophil count > 1.5 ×109/L
* Platelet count ≥ 50.0 ×109/L
* Total bilirubin < 51 μmol/L
* Alanine transaminase (ALT) and aminotransferase (AST) < 5 x upper limit of normal
* Albumin > 28 g/L
* Prothrombin time (PT)-international normalized ratio (INR) < 2.3, or PT < 6 seconds above control
* Serum creatinine < 110 μmol/L
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

* A history of liver decompensation, such as refractory ascites, gastrointestinal bleeding, or hepatic encephalopathy; Uncontrolled complications, including but not limited to: Persistent or activity (except the HBV and HCV) infection, symptoms of congestive heart failure and uncontrolled diabetes, uncontrolled hypertension, unstable angina, uncontrolled arrhythmias, active ILD, severe chronic GI disease accompanied by diarrhea, or compliance with requirements may limit the research, resulted in significant increase risk of AE or influence Subjects provided psychiatric/social problem status on their ability to provide written informed consent. A history of active primary immunodeficiency or human immunodeficiency virus; Active or previous records of autoimmune disease or inflammatory diseases, including inflammatory bowel disease (e.g., colitis or Crohn's disease], diverticulitis, except [diverticulosis], systemic lupus erythematosus (SLE), sarcoidosis syndrome or Wegener syndrome (e.g., granulomatous vasculitis, gray's disease, rheumatoid arthritis, the pituitary gland inflammation and uveitis]).
* Known to produce allergic or hypersensitive reactions to any study drug or any excipient thereof;
* Significant clinical gastrointestinal bleeding or a potential risk of bleeding was identified by the investigator during the 30 days prior to study entry.
* Tumors of the central nervous system, including metastatic brain tumors;
* Pregnant women or breast-feeding patients;
* Complicated with other malignant tumors:
* Malignant tumors that have been treated for therapeutic purposes, have no known active disease for 5 years prior to the first administration of the study drug, and have a low potential risk of recurrence.
* Fully treated non-melanoma skin cancer or malignant freckle moles with no evidence of disease.
* Fully treated carcinoma in situ without evidence of disease.
* Prior to the initial dosing of the study drug, they had received anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapy.
* Has received anti-tumor system therapy for HCC. Non-anti-tumor purpose combined hormone therapy (e.g., hormone replacement therapy) is excluded.
* Is currently using, or has used an immunosuppressive drug within 14 days prior to the first dose of the investigational drug. This standard has the following exceptions:
* intranasal, inhaled, topical or topical steroids. (e.g., intraarticular)
* Systemic corticosteroid therapy not exceeding 10 mg/ day of prednisone or its physiological equivalent as a prophylactic use of steroids for hypersensitivity. (e.g., CT scan pretherapy medication)
* Steroids as a prophylactic for allergic reactions.
* A live attenuated vaccine was administered within 30 days prior to the first administration of the study drug. Note: If enrolled, patients shall not receive live attenuated vaccine within 30 days of receiving study drug therapy and after the last administration of study drug.
* Uncontrolled hypertension: systolic pressure ≥ 160 mmHg or diastolic pressure ≥ 100 mmHg despite anti-hypertension medications ≤ 28 days before randomization or first dose of drug.
* Pregnant or lactating women, or fertile men or women who do not want to use high-efficiency contraceptives, 6 months after the last dosing of study treatment, from screening to study treatment. Based on the patient's preferred and customary lifestyle, abstinence during treatment and washout is an acceptable contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sequential and maintenance therapy of Regorafenib plus ICIs in andvanced HCC patients who have completed standard HAIC.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-16 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2-years Followed up
  Absence of death of any cause
Progress Free Survival | 2-years Followed up
  Absence of disease progression other than death

SECONDARY OUTCOMES:
Tumor local control | 2-years Followed up
  Absence of regrowth inside the treated lesion
Adverse Events (AEs) | 2-years Followed up
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0
Tumor Response | 2-years Followed up
  Tumor response to Regorafenib Combined With ICIs according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, M.D. & Ph.D., Principal Investigator — Department of Minimally Invasive and Interventional Radiology, Liver Cancer
Locations (2):
- China (2):
  - Department of Minimally Invasive and Interventional Radiology, Liver Cancer Study and Service Group, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lyu N, Wang X, Li JB, Lai JF, Chen QF, Li SL, Deng HJ, He M, Mu LW, Zhao M. Arterial Chemotherapy of Oxaliplatin Plus Fluorouracil Versus Sorafenib in Advanced Hepatocellular Carcinoma: A Biomolecular Exploratory, Randomized, Phase III Trial (FOHAIC-1). J Clin Oncol. 2022 Feb 10;40(5):468-480. doi: 10.1200/JCO.21.01963. Epub 2021 Dec 14. PMID 34905388
- [Background] Lyu N, Kong Y, Mu L, Lin Y, Li J, Liu Y, Zhang Z, Zheng L, Deng H, Li S, Xie Q, Guo R, Shi M, Xu L, Cai X, Wu P, Zhao M. Hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin vs. sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):60-69. doi: 10.1016/j.jhep.2018.02.008. Epub 2018 Feb 20. PMID 29471013
- [Background] Lyu N, Lin Y, Kong Y, Zhang Z, Liu L, Zheng L, Mu L, Wang J, Li X, Pan T, Xie Q, Liu Y, Lin A, Wu P, Zhao M. FOXAI: a phase II trial evaluating the efficacy and safety of hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin for advanced hepatocellular carcinoma. Gut. 2018 Feb;67(2):395-396. doi: 10.1136/gutjnl-2017-314138. Epub 2017 Jun 7. No abstract available. PMID 28592441